CLINICAL TRIAL: NCT02429947
Title: An Analysis of the Symptomatic Domains Most Relevant to Charcot Marie Tooth Neuropathy (CMT) Patients
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: University of Rochester (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: INC6606; 5U54NS064808-07 (NIH); INC6606 (Other: Inherited Neuropathies Consortium)
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Charcot Marie Tooth Disease (CMT); Hereditary Sensory and Motor Neuropathy; Nerve Compression Syndromes; Tooth Diseases; Congenital Abnormalities; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System
Keywords: Charcot Marie Tooth disease; CMT; HMSN; HMN; HSN
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Hereditary Sensory and Motor Neuropathy; Nerve Compression Syndromes; Tooth Diseases; Congenital Abnormalities; Genetic Diseases, Inborn; Heredodegenerative Disorders, Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INC Contact Registry Participants: Adult CMT patients who have self-registered at the Inherited Neuropathies Consortium (INC) Contact Registry, a web-based contact registry developed and supported by the Data Management and Coordinating Center (DMCC) for the Rare Diseases Clinical Research Consortium (RDCRN), located at the University of South Florida.

SUMMARY:
The purpose of this study is to identify the issues that have greatest impact on QOL for patients with Charcot Marie Tooth (CMT) Disease. Patients who have -registered in the Inherited Neuropathies Consortium Contact Registry will be invited to participate.

DETAILED DESCRIPTION:
The protocol consists of two anonymous surveys. The first large scale survey is designed to identify items that best reflect the issues and symptoms with high impact upon QOL in CMT. A second brief survey focuses on the frequency and impact of muscle cramps on QOL in adult CMT. The surveys will be distributed via an online link to all adult CMT patients self-registered with the RDCRN contact registry. Those who complete the first two surveys will be requested to complete only the second brief survey on muscle cramps again 3 weeks after completing it the first time. Those who complete the brief muscle cramps survey a second time will be requested to complete it again 5 weeks later to assess variability in occurrence of muscle cramps.

The first large scale survey to identify items that best reflect the issues and symptoms with high impact upon QOL in CMT will be sent out in a second wave. This second wave will only contain the QOL survey and not the muscle cramp survey. The QOL survey will be distributed via an online link to three populations: adult CMT patients self-registered with the INC (RDCRN) Contact Registry who had not been registered at the time of the first enrollment period, adult patients who had been registered at the time of the first enrollment period and had received the survey, but had not returned it, and patients who were registered, but were under age 18 at the time of the first enrollment period and have turned 18 by the time of the second enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CMT that are 18 years or older and have joined the INC RDCRN Contact Registry.

Exclusion Criteria:

* Does not have CMT.
* Does not read or speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CMT, 18 years or older, who have joined the Inherited Neuropathies Consortium RDCRN Contact Registry.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants affected by specific symptoms of CMT. | 1 year
  The percentage of subjects within the sample who have reported experience with the symptom will be calculated.

SECONDARY OUTCOMES:
Severity of impact of each identified symptom of CMT | 1 year
  The symptoms will be rank ordered with symptoms that affect life severely receiving the highest rank.

CONTACTS AND LOCATIONS:
Overall Officials: David Herrmann, MBBCh, Study Chair — University of Rochester
Locations (1):
- RDCRN Data Management and Coordinating Center , Epidemiology Center; University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No